CLINICAL TRIAL: NCT00993798
Title: An International, Randomised, Double Blinded, Multi-centre, Active- and Placebo-controlled Dose Response Trial to Evaluate the Efficacy and Safety of SABER-Bupivacaine for Postoperative Pain Control in Patients Following Arthroscopic Shoulder Surgery
Brief Title: An International Trial to Evaluate the Efficacy and Safety of SABER®-Bupivacaine for Postoperative Pain Control in Patients Following Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BU-002-IM
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Post operative pain; Local anaesthesia; Postoperative pain after arthroscopic shoulder surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SABER-Bupivacaine Treatment 1a (Experimental): double-blind
  Interventions: Drug: SABER-Bupivacaine Treatment 1a
- Placebo SABER-Bupivacaine Treatment 1b (Placebo Comparator): double-blind
  Interventions: Drug: Placebo SABER-Bupivacaine Treatment 1b
- Bupivacaine HCl Treatment 1c (Active Comparator): double-blind
  Interventions: Drug: Bupivacaine HCl Treatment 1c
- SABER-Bupivacaine Treatment 2a (Experimental): double-blind
  Interventions: Drug: SABER-Bupivacaine Treatment 2a
- Placebo SABER-Bupivacaine Treatment 2b (Placebo Comparator): double-blind
  Interventions: Drug: Placebo SABER-Bupivacaine Treatment 2b
- Bupivacaine HCl Treatment 2c (Active Comparator): double-blind
  Interventions: Drug: Bupivacaine HCl Treatment 2c

INTERVENTIONS:
Drug: SABER-Bupivacaine Treatment 1a — 5.0 ml
  Other Names: POSIMIR® bupivacaine solution
  Arms: SABER-Bupivacaine Treatment 1a
Drug: Placebo SABER-Bupivacaine Treatment 1b — 5.0 ml
  Arms: Placebo SABER-Bupivacaine Treatment 1b
Drug: Bupivacaine HCl Treatment 1c — 20.0 ml
  Arms: Bupivacaine HCl Treatment 1c
Drug: SABER-Bupivacaine Treatment 2a — 7.5 ml
  Arms: SABER-Bupivacaine Treatment 2a
Drug: Placebo SABER-Bupivacaine Treatment 2b — 7.5 ml
  Arms: Placebo SABER-Bupivacaine Treatment 2b
Drug: Bupivacaine HCl Treatment 2c — 20.0 ml
  Arms: Bupivacaine HCl Treatment 2c

SUMMARY:
The objective is to identify the optimal dose of SABER-Bupivacaine for postoperative pain control in patients undergoing elective arthroscopic shoulder surgery on the basis of pharmacokinetics, efficacy and safety evaluations. The study duration consists of a screening period up to 14 days and a treatment period 14 days with a long term follow up visit at 6 months. The study will provide further data on safety.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial impingement syndrome
* MRI with intact rotator cuff
* Patients suitable for general anaesthesia

Exclusion Criteria:

* Known major joint trauma, infection, avascular necrosis, chronic dislocation, inflammatory or degenerative glenohumeral arthropathy, glenohumeral arthritis, frozen shoulder or previous surgery of the affected shoulder
* Abnormal ECG
* Prolonged QT syndrome
* Current or regular use of analgesic medication for other indication(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (9):
- Austria (2):
  - Nycomed Investigational Site, Graz
  - Nycomed Investigational Site, Vienna
- Germany (3):
  - Nycomed Investigational Site, Berlin
  - Nycomed Investigational Site, Dresden
  - Nycomed Investigational Site, Marburg
- Latvia (2):
  - Nycomed Investigational Site, Riga
  - Nycomed Investigational Site, Valmiera
- Nycomed Investigational Site, Lodz, Poland
- Nycomed Investigational Site, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter, randomized, double-blind, parallel-group, placebo- and active-controlled study in adult subjects undergoing elective arthroscopic subacromial decompression.
Groups:
- SABER-Bupivacaine 5 mL; SABER-placebo 5 mL: 5 mL, single dose instilled subacromially
- Bupivacaine HCl 0.25% 20 mL: 0.25% 20 mL, single dose instilled subacromially
- SABER- Placebo 7.5 mL; SABER-Bupivacaine 7.5 mL: 7.5 mL, single dose instilled subacromially. This arm was never pursued.
Period: Overall Study
Arm/Group | SABER-Bupivacaine 5 mL | SABER-placebo 5 mL | Bupivacaine HCl 0.25% 20 mL | SABER- Placebo 7.5 mL | SABER-Bupivacaine 7.5 mL
Started | 53 | 25 | 29 | 0 | 0
Completed | 53 | 25 | 29 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SABER-Bupivacaine; SABER-placebo: 5 mL, single dose instilled subacromially
- Bupivacaine HCl: 0.25% 20 mL, single dose instilled subacromially
- Total: Total of all reporting groups
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl | Total
Number analyzed (Participants) | 53 | 25 | 29 | 107
Age, Continuous [Mean (Full Range); unit: years] | 50.1 [28 to 70] | 48.6 [24 to 63] | 51.6 [21 to 70] | 50.2 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 17 | 64
  Male | 20 | 11 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (PI)
Description: Mean pain intensity on movement AUC (time-normalized AUC) during the period 0-3 days after surgery. Pain intensity was assessed with a standard 0 to 10 numeric rating scale (NRS), where no pain at all was rated as 0 and the worst pain imaginable was rated as 10. The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 0-3 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (time-normalized AUC)
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 53 | 25 | 29
score on a scale (time-normalized AUC) | 5.16 (1.94) | 6.43 (1.77) | 5.16 (2.38)
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.012, t-test in ANOVA model; LS Mean Difference = -1.27, 95% CI 2-sided [-2.25 to -0.28], Standard Deviation 0.50

2. Primary Outcome: Supplemental Opioid Use
Description: Cumulative IV morphine-equivalent dose of opioid rescue medication
Time Frame: 0-3 days after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 53 | 25 | 29
mg | 4.0 [0.0 to 15.0] | 12.0 [4.0 to 36.0] | 8.0 [0.0 to 16.0]
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -8.0, 95% CI 2-sided [-12.0 to 0.0]

3. Secondary Outcome: Time to First Opioid Rescue Medication Usage
Time Frame: 0-14 days after surgery
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 53 | 25 | 29
hours | 12.4 [1.2 to NA] — The confidence interval is for a median estimated by a Kaplan-Meier curve. There were too few events overall to estimate an upper endpoint for this interval. | 1.2 [0.7 to 1.5] | 1.4 [1.0 to 4.1]
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.014, Log Rank

4. Secondary Outcome: Opioid Related Side Effects
Description: Opioid-related side effects were recorded 0-7 days after surgery. The Opioid-Related Symptom Distress Scale (OR-SDS) is a composite score computed from a questionnaire containing frequent opioid-related symptoms (Fatigue, Drowsiness, Inability to concentrate, Nausea, Dizziness, Constipation, Itching, Difficulty with urination, Confusion, Retching/vomiting). For each symptom, patients assigned integer scores to assess severity (none=0 to very severe=4), bothersomeness (none=0 to very much=5), and frequency (none=0 to almost constantly=4); patients reported number of Retching/vomiting episodes (none=0, 1-2 episodes=1, 3-4 episodes=2, 5-6 episodes=3, >6 episodes=4).
  On each day (Day 0-7), the score for each symptom was the mean of the three component scores, and the OR-SDS score was the overall mean of the 10 symptom scores, (values from 0 to 4; larger outcomes are worse). The mean of the daily OR-SDS score from Day 0 to 7 gave the overall OR-SDS Score.
Time Frame: 0-7 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 37 | 21 | 23
score on a scale | 0.22 (0.35) | 0.22 (0.24) | 0.25 (0.24)
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.773, ANOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.18 to 0.14], Standard Deviation 0.08

ADVERSE EVENTS:
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/25 | 4/29
Other Adverse Events (participants affected / at risk) | 12/53 | 6/25 | 6/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (N=53) | SABER-placebo (N=25) | Bupivacaine HCl (N=29)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drug intolerance (General disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tongue paralysis (Nervous system disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (N=53) | SABER-placebo (N=25) | Bupivacaine HCl (N=29)
Headache (Nervous system disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
ALT increased (Investigations) | 1 | 2 | 0
ECG T wave abnormal (Investigations) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes